CLINICAL TRIAL: NCT06988397
Title: Food Type and Physical Activity Influence on Gastric Emptying Time Assessed by Ultrasound in Healthy Volunteers
Brief Title: Stomach Processing and Emptying Evaluation With Diet and Ultrasound
Acronym: SPEED-US
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Medical University of Warsaw (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Diagnostic
Other Study IDs: KB/6/2025
Record Dates: First submitted 2025-04-17; First posted 2025-05-23 (Actual); Last update posted 2025-05-23 (Actual); Status verified 2025-05

CONDITIONS: Gastric Emptying; Preoperative Risk Assessment; Healthy Volunteer Study
Keywords: Gastric emptying; Gastric volume; Ultrasound; Gastric POCUS

STUDY DESIGN:
Who Masked: Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Gastric Ultrasound in Participants Consuming Different Meal Types with Physical Acivity (Experimental): Participants assigned to this arm will undergo an initial gastric ultrasound to confirm fasting status. They will then consume one of three types of meals: vegetable-based, meat-based, or dairy-based. A gastric ultrasound will be performed 15 minutes after meal ingestion. This will be followed by standardized physical activity (walking a predefined distance). Subsequent gastric ultrasound assessments will be performed at 3 hours and 6 hours post-meal, each followed by the same standardized physical activity. The purpose is to evaluate the impact of food type and intermittent physical activity on gastric emptying, as assessed by ultrasound.
  Interventions: Behavioral: Physical activity after different type of meals
- Gastric Ultrasound in Participants Consuming Different Meal Types with Subsequent Rest (No Intervention): Participants in this arm will first undergo a baseline gastric ultrasound to confirm fasting status. They will then consume one of three types of meals: vegetable-based, meat-based, or dairy-based. Gastric ultrasound will be performed 15 minutes after meal ingestion. Unlike the other arm, participants in this group will remain at rest throughout the study period and will not perform any physical activity. Additional gastric ultrasound assessments will be performed at 3 hours and 6 hours post-meal, with participants remaining sedentary between each measurement. This arm will serve to assess the isolated effect of food type on gastric emptying over time without the influence of physical activity.

INTERVENTIONS:
Behavioral: Physical activity after different type of meals — Standardized physical activity (walking) after consuming one of three meal types (vegetable-based, meat-based, dairy-based). Ultrasound of gastric volume will be performed at 3 and 6 hour between walking sessions.
  Arms: Gastric Ultrasound in Participants Consuming Different Meal Types with Physical Acivity

SUMMARY:
Gastric content is a key risk factor for aspiration during anesthesia. Although standard fasting times are recommended, various factors-including GLP-1 receptor agonists,-can delay gastric emptying. Gastric ultrasound enables real-time, non-invasive assessment of gastric volume and can help tailor perioperative management. The aim of this study explores the effects of different meal types and physical activity on gastric emptying in healthy individuals.

DETAILED DESCRIPTION:
Pulmonary aspiration of gastric contents is a serious and potentially life-threatening complication of anesthesia. Despite adherence to preoperative fasting guidelines issued by the American Society of Anesthesiologists (ASA), certain medical conditions-such as diabetes mellitus-or medications like GLP-1 receptor agonists may significantly delay gastric emptying beyond standard expectations. This creates a need for individualized assessment of gastric contents prior to anesthesia, especially in patients considered at increased risk.

Gastric ultrasound is a non-invasive, point-of-care technique that allows for real-time assessment of gastric volume and content. It may provide a more reliable indicator of aspiration risk than fasting time alone.

This randomized, prospective study aims to evaluate the effects of different types of meals and physical activity levels on gastric emptying time in healthy adult volunteers, using ultrasound-based measurement of the gastric antrum.

Sixty participants aged 18-40 years will be recruited via registration forms provided by the study team. Each participant will provide written informed consent, including acknowledgment of potential food allergens present in the study meals. The day prior to each session, participants will receive a phone call to remind them of dietary restrictions: no clear liquids for 2 hours, no solid foods for 6 hours, and no fatty meals for 8 hours before the study.

Each participant will take part in two separate sessions, conducted on different days. On both days, the participant will arrive fasting and undergo a baseline gastric ultrasound to confirm an empty stomach. If gastric content is detected, the session will be rescheduled.

Participants will be randomly assigned (via computer-generated allocation) to one of three meal groups: high-fat, dairy-based, or fruit/vegetable. Meals will be standardized in volume and composition within each group. The examiner performing the ultrasound will be blinded to the meal group allocation.

In each session, participants will consume the assigned meal within 10 minutes. Gastric ultrasound measurements will be performed at 15 minutes, 3 hours, and 6 hours post-meal. On one of the days, participants will remain in a resting position between measurements. On the other day, participants will walk at a moderate pace for 30 minutes between each measurement interval (i.e., between 0-3 hours and 3-6 hours post-meal). The order of active vs. resting day will be randomized and counterbalanced across participants.

Ultrasound will be performed in the right lateral decubitus position using a convex transducer (2-8 MHz) with an abdominal preset. The antral cross-sectional area (CSA) will be measured using standard landmarks (aorta, SMA, left lobe of liver), and gastric volume will be estimated using a validated formula:

GV = 27.0 + 14.6 × right lateral CSA (cm²) - 1.28 × age (years).

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 40 years
* Ability and willingness to provide written informed consent
* Agreement to comply with study procedures, including pre-study dietary restrictions
* No history of gastrointestinal disease
* No recent abdominal surgery

Exclusion Criteria:

* Lack of informed consent
* Allergy or intolerance to any of the foods used in the study meals
* Medical conditions known to delay gastric emptying, including:
* Obesity (BMI > 30 kg/m²)
* Diabetes mellitus
* Gastroesophageal reflux disease (GERD)
* Hiatal hernia
* Bowel obstruction
* Tube feeding
* Active gastrointestinal disease
* History of gastrointestinal surgery
* Current pregnancy or breastfeeding
* Use of medications affecting gastric motility (e.g., opioids, anticholinergics, GLP-1 receptor agonists)
* Neuromuscular disorders impairing ability to remain in supine position for 6 hours or to walk for 30 minutes

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 60 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2026-05-01 (Estimated); Study Completion 2026-06-01 (Estimated)

PRIMARY OUTCOMES:
Time to ultrasonographic signs of an empty stomach | after 15 minutes, 3 hours and 6 hours post-meal
  Time (in hours) required to reach a gastric ultrasound profile consistent with an empty stomach (defined individually based on baseline fasting scan), depending on physical activity and meal type

SECONDARY OUTCOMES:
Antral cross-sectional area (CSA) | at 15 minutes, 3 hours, and 6 hours post-meal
  Changes in CSA (cm²)
Estimated gastric volume (GV) | At 15 minutes, 3 hours, and 6 hours post-meal
  Calculated from CSA and age using validated formula

CONTACTS AND LOCATIONS:
Overall Officials: Mateusz Zawadka, Principal Investigator — 2nd Department of Anesthesiology and Intensive Care, Medical University of Warsaw, Poland
Locations (1):
- Medical University of Warsaw, Warsaw, Masovian Voivodeship, Poland

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Van de Putte P, Perlas A. Ultrasound assessment of gastric content and volume. Br J Anaesth. 2014 Jul;113(1):12-22. doi: 10.1093/bja/aeu151. Epub 2014 Jun 3. PMID 24893784
- [Background] Bolondi L, Bortolotti M, Santi V, Calletti T, Gaiani S, Labo G. Measurement of gastric emptying time by real-time ultrasonography. Gastroenterology. 1985 Oct;89(4):752-9. doi: 10.1016/0016-5085(85)90569-4. PMID 3896910
- [Background] Perlas A, Chan VW, Lupu CM, Mitsakakis N, Hanbidge A. Ultrasound assessment of gastric content and volume. Anesthesiology. 2009 Jul;111(1):82-9. doi: 10.1097/ALN.0b013e3181a97250. PMID 19512861
- [Background] Sumpelmann AE, Sumpelmann R, Lorenz M, Eberwien I, Dennhardt N, Boethig D, Russo SG. Ultrasound assessment of gastric emptying after breakfast in healthy preschool children. Paediatr Anaesth. 2017 Aug;27(8):816-820. doi: 10.1111/pan.13172. Epub 2017 Jul 4. PMID 28675504
- [Background] Pimenta GP, de Aguilar-Nascimento JE. Prolonged preoperative fasting in elective surgical patients: why should we reduce it? Nutr Clin Pract. 2014 Feb;29(1):22-8. doi: 10.1177/0884533613514277. Epub 2013 Dec 11. PMID 24336400
- [Background] Practice Guidelines for Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration: Application to Healthy Patients Undergoing Elective Procedures: An Updated Report by the American Society of Anesthesiologists Task Force on Preoperative Fasting and the Use of Pharmacologic Agents to Reduce the Risk of Pulmonary Aspiration. Anesthesiology. 2017 Mar;126(3):376-393. doi: 10.1097/ALN.0000000000001452. No abstract available. PMID 28045707